CLINICAL TRIAL: NCT00274443
Title: An Open -Label, Phase II Trial of Increasing Doses of ABI-007 and Carboplatin in Patients With Advanced Non Small Cell Lung Cancer (NSCLC)
Brief Title: An Open Label Study in Patients With Advanced NSCLC With ABI-007(Abraxane) in Combination With Carboplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA028
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-007 and Carboplatin (Experimental): ABI-007 and Carboplatin in patients with Advanced Non-Small Cell Lung Cancer.
  Interventions: Drug: ABI-007 (Abraxane) and Carboplatin

INTERVENTIONS:
Drug: ABI-007 (Abraxane) and Carboplatin — ABI-007 plus Carboplatin will be administered intravenously over 30 minutes in cycles of 3 weeks

SUMMARY:
This is an open-label dose escalation trial using ABI-007 plus carboplatin.

DETAILED DESCRIPTION:
This is a multicenter study conducted at study sites in Russia and the Ukraine where various doses of ABI-007 (Abraxane) will be given in combination with carboplatin to patients with non-small cell lung cancer to determine the recommended dose and schedule for this combination therapy for Phase III trials. The primary objective of this study is to obtain preliminary information on the antitumor activity and adverse events of ABI-007 in combination with carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC Stage IIIB with pleural effusion or evidence of inoperable local recurrence or metastasis (Stage IV).
* Male or non-pregnant and non-lactating female, and ≥ 18 years of age. ( )If a female patient is of child-bearing potential, as evidenced by regular menstrual periods, she must have a negative serum pregnancy test (β-hCG) documented within 72 hours of the first administration of study drug. ( )If sexually active, the patient must agree to utilize contraception considered adequate and appropriate by the investigator.
* No other current active malignancy.
* Measurable disease
* Patients must have received no prior therapy for the treatment of metastatic disease.
* Patient has the following blood counts at baseline:

( ) ANC ≥ 1.5 x 109/L; ( ) platelets ≥ 100 x 109/L; ( ) Hgb ≥ 9 g/dL.

* Patient has the following blood chemistry levels at baseline:

( ) AST (SGOT), ALT (SGPT) ≤ 1.5x upper limit of normal range (ULN); ( ) total bilirubin NORMAL; ( ) creatinine ≤ 1.5 mg/dL.

* Expected survival of > 12 weeks.
* ECOG performance status 0 or 1.
* Patient or his/her legally authorized representative or guardian has been informed about the nature of the study, and has agreed to participate in the study, and signed the Informed Consent form prior to participation in any study-related activities.

Exclusion Criteria:

* Evidence of active brain metastases, including leptomeningeal involvement. Prior evidence of brain metastasis permitted only if treated and stable off therapy for at least 1 month.
* The only evidence of metastasis is bone metastases or other nonmeasurable disease.
* Patient has pre-existing peripheral neuropathy of grade 2, 3, or 4.
* Patient received radiotherapy in last 4 weeks, except if to a non-target lesion only. Prior radiation to a target lesion is permitted only if there has been clear progression of the lesion since radiation was completed.
* Patient has a clinically significant concurrent illness.
* Patient is, in the investigator's opinion, unlikely to be able to complete the study through the End of Study visit.
* Patient has received treatment with any other cytotoxic chemotherapeutic agent or investigational drug within the previous 4 weeks;
* Patient has a history of allergy or hypersensitivity to the study drug.
* Patient has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the patient to receive an experimental research drug.
* Patient is enrolled in any other clinical protocol or investigational trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2007-06-01 (Actual)

PRIMARY OUTCOMES:
Safety Outcomes: incidence of treatment emergent adverse events. | Treatment duration
Efficacy Outcomes: percentage of patients who achieve an objective confirmed complete or partial overall antitumor response | Treatment duration

CONTACTS AND LOCATIONS:
Locations (1):
- Study Sites in Russia, Saint Petersburg, Sankt-Peterburg, Russia

REFERENCES:
- [Background] Socinski MA, Manikhas GM, Stroyakovsky DL, Makhson AN, Cheporov SV, Orlov SV, Yablonsky PK, Bhar P, Iglesias J. A dose finding study of weekly and every-3-week nab-Paclitaxel followed by carboplatin as first-line therapy in patients with advanced non-small cell lung cancer. J Thorac Oncol. 2010 Jun;5(6):852-61. doi: 10.1097/jto.0b013e3181d5e39e. PMID 20521351